CLINICAL TRIAL: NCT02617654
Title: A Randomized, Double-blinded Placebo-controlled, Paralleled Designed, Investigator Sponsored Study of the Effect of the GLP-1 Receptor Agonist Liraglutide on Beta-cell Function in C-peptide Positive Type 1 Diabetic Patients
Brief Title: Liraglutide Effect on Beta-cell Function in C-peptide Positive Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Per-Ola Carlsson (Other)
Responsible Party: Sponsor-Investigator, Per-Ola Carlsson, Professor, senior consultant, Uppsala University Hospital
Organization: Uppsala University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U1111-1166-6923
Record Dates: First submitted 2015-11-20; First posted 2015-12-01 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide treatment (Active Comparator): Liraglutide treatment in the dose of 1.8 mg daily for 52 weeks
  Interventions: Drug: Liraglutide
- Placebo treatment (Placebo Comparator): Treatment with placebo once daily for 52 weeks
  Interventions: Drug: Placebo for liraglutide

INTERVENTIONS:
Drug: Liraglutide — Treatment with liraglutide for 52 weeks
  Arms: Liraglutide treatment
Drug: Placebo for liraglutide — Placebo for liraglutide. Treatment once daily for 52 weeks
  Arms: Placebo treatment

SUMMARY:
Recent studies show that many Type 1 diabetes patients have remaining endogenous insulin production, albeit at low levels. Finding means to increase this production would be of tremendous interest, since residual C-peptide concentrations >0.1 nmol/l previously have been shown to markedly lower HbA1c, decrease blood glucose fluctuations and diminish the risk of ketoacidosis. It also substantially reduces the risks of severe hypoglycemic events and late complications. Liraglutide may through its incretin effect directly potentiate beta-cell function, but also holds the potential to be mitogenic for these cells.

The hypothesis of the present trial is that treatment with liraglutide will not only have a direct effect on beta-cell function, which is more or less immediately observed, but also progressively improve C-peptide concentrations over time.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for participation of the study, given before undergoing any study-specific procedures.
2. 18-30 years of age (age interval inclusive of both the ends). Both males and females are eligible for the study
3. Clinical diagnose of T1D
4. Five or more years duration of disease
5. HbA1C between 45 and 75 mmol/mol
6. Fasting plasma C-peptide concentration >1.5 pmol/l.

Exclusion Criteria:

1. Inability to provide informed consent
2. Mental incapacity
3. Unwillingness or language barrier precluding adequate understanding or cooperation
4. Ongoing or planned pregnancy within the next 12 months
5. Inadequate or no use of contraceptives
6. Ongoing breast feeding
7. Known sight-threatening retinopathy
8. Creatinine clearance <60 ml/min
9. Life-threatening cardiovascular disease
10. History of drug/alcohol abuse
11. Known or suspected allergy to trial product or related product
12. Recurrent assisted hypoglycemias
13. Taking oral anti-diabetic therapies or any other concomitant medication which may interfere with glucose regulation other than insulin
14. Uncontrolled hypertension (180/105 mmHg or above)
15. History of acute or chronic pancreatitis
16. Personal or family history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma (FMTC)
17. Personal history of non-familial medullary thyroid carcinoma.
18. Any condition that the investigator or sponsor feel would interfere with trial participation or evaluation of results

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-11; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
The effect of 52 weeks of treatment with liraglutide 1.8 mg/day, compared to placebo, on stimulated C-peptide concentrations in patients with long-standing type 1 diabetes and residual insulin production | 52 weeks
  The Area Under the Curve (AUC) change in plasma C-peptide concentration in response to a standardized mixed meal tolerance test (MMTT) during one year of liraglutide treatment (1.8 mg/day)

SECONDARY OUTCOMES:
Change in C-peptide between 6 and 52 weeks of study | 52 weeks
  ∆- change in C-peptide AUC between the MMTT after one year and that after 6 weeks of treatment
Change in C-peptide between after and prior to treatment with liraglutide 1.8 mg | 52 weeks
  ∆-change in C-peptide AUC between the MMTT three months after cessation of treatment and that after the run-in period
Change in HbA1c between before and at end of liraglutide (1.8 mg) treatment | 52 weeks
  ∆- change in HbA1c between after one year and after the run-in period.
Change in HbA1c between 6 and 52 weeks of study | 52 weeks
  ∆- change in HbA1c between after one year and after 6 weeks of treatment
Change in HbA1c between after and prior to treatment with liraglutide 1.8 mg | 52 weeks
  ∆- change in HbA1c between three months after the cessation of treatment and after the run-in period.
Change in insulin doses between before and at end of liraglutide (1.8 mg) treatment | 52 weeks
  ∆- change in exogenous insulin doses between after one year and after the run-in period.
Change in insulin doses between 6 and 52 weeks of study | 52 weeks
  ∆- change in exogenous insulin doses between after one year and after 6 weeks of treatment
Change in insulin doses between after and prior to treatment with liraglutide 1.8 mg | 52 weeks
  ∆- change in exogenous insulin doses between three months after the cessation of treatment and after the run-in period.
Change in glucose variability between before and at end of liraglutide (1.8 mg) treatment | 52 weeks
  ∆- change in glucose variability between after one year and after the run-in period.
Change in glucose variability between 6 and 52 weeks of study | 52 weeks
  ∆- change in glucose variability between after one year and after 6 weeks of treatment
Change in glucose variability between after and prior to treatment with liraglutide 1.8 mg | 52 weeks
  ∆- change in glucose variability between three months after the cessation of treatment and after the run-in period.
Change in hypoglycemia frequency between before and at end of liraglutide (1.8 mg) treatment | 52 weeks
  ∆- change in hypoglycemia frequency (measured plasma glucose levels < 3 mmol/l or assisted hypoglycemia during a one week period) between one year and after the run-in period.
Change in hypoglycemia frequency between 6 and 52 weeks of study | 52 weeks
  ∆- change in hypoglycemia frequency (measured plasma glucose levels < 3 mmol/l or assisted hypoglycemia during a one week period) after one year and after 6 weeks of treatment
Change in hypoglycemia frequency between after and prior to treatment with liraglutide 1.8 mg | 52 weeks
  ∆- change in hypoglycemia frequency (measured plasma glucose levels < 3 mmol/l or assisted hypoglycemia during a one week period) between three months after the cessation of treatment and after the run-in period.
Change in Quality of Life (QoL) between before and at end of liraglutide (1.8 mg) | 52 weeks
  ∆- change in assessment of QoL between after one year and after the run-in period.
Change in QoL between 6 and 52 weeks of study | 52 weeks
  ∆- change in assessment of QoL between after one year and after 6 weeks of treatment
Change in QoL between after and prior to treatment with liraglutide | 52 weeks
  ∆- change in assessment of QoL between three months after the cessation of treatment and after the run-in period.

CONTACTS AND LOCATIONS:
Overall Officials: Per-Ola Carlsson, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden